CLINICAL TRIAL: NCT05438758
Title: Phase 2, Controlled, Single-Blind, 3-Month Extension Study For Participants Originally Diagnosed With Treatment Resistant Major Depressive Disorder (TRD) Who Complete Study ZYL-730-01 With, or Without, Almond Therapy
Brief Title: Repeated Intranasal Esketamine Plus Almond Therapy in Participants With Treatment Resistant Depressive Disorder - 3 Month Extension Study
Acronym: ZYL-730-02
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn by Sponsor
Sponsor: Zylorion Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HREBA-CTC-22-0066
Record Dates: First submitted 2022-06-24; First posted 2022-06-30 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Treatment Resistant Major Depressive Disorder
MeSH Terms: interventions — Esketamine; Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants who have received Almond Therapy in study ZYL-730-01 will continue to have this in the extension study Participants who received Treatment as Usual in study ZYL-730-02 will continue to have this in the extension study.
Who Masked: Outcomes Assessor
Masking Description: The independent trained individual will not be aware of which treatment arm the participant is in. The Montgomery Asberg Depression Rating Scale (MADRS) assessor will have no other contact with participant apart from remotely assessing the MADRS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal Esketamine with Addition of Almond TherapyTM (Other): Intranasal Esketamine - Dose of 56 mg or 84 mg once a week for 4 weeks followed by 56 mg or 84 mg once every two weeks for 8 weeks.
  Interventions: Behavioral: Almond Therapy; Drug: Intranasal ketamine (Esketamine)
- Intranasal Esketamine with Treatment as Usual (Other): Intranasal Esketamine - Dose of 56 mg or 84 mg once a week for 4 weeks followed by 56 mg or 84 mg once every two weeks for 8 weeks.
  Interventions: Drug: Intranasal ketamine (Esketamine); Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Almond Therapy — Participants will receive 12 remote session conducted by video or phone. Therapy sessions consist of modules selected using a shared decision making process, tailored so that it is personally meaningful to each participants. Participants will also receive supportive text messages on selective days over the 3 months.
  Arms: Intranasal Esketamine with Addition of Almond TherapyTM
Drug: Intranasal ketamine (Esketamine) — Participants will receive 56 mg or 84 mg once a week for 4 weeks followed by 56 mg or 84 mg once every two weeks for 8 weeks
Behavioral: Treatment as Usual — Participants will continue to received the therapy that their treating physician felt was appropriate at the time of enrolment in the study. These can include cognitive behavioural therapy, supportive psychotherapy or mindfulness, support groups, physical activity or relaxation.
  Arms: Intranasal Esketamine with Treatment as Usual

SUMMARY:
The purpose of this study is to determine if any improvements in depressive symptoms are maintained in the medium and longer-term (up to 3 months)

DETAILED DESCRIPTION:
The duration of the study is 3 months

Participants enrolled in the Almond Therapy group will have up to 9 in person visits, including the baseline visits, participants will receive Esketamine on 8 of these visits. There are 12 remote therapy sessions conducted via telephone or video, participants will also receive supportive text messages. In addition, participants will have 4 telephone calls from an independent assessor to ask questions about their mental health (MADRS).

Participants enrolled in the Treatment as Usual group will have up to 9 in person visits, including the baseline visits, participants will receive Esketamine on 8 of these visits. Participants will continue to receive the therapy their treating physician felt was appropriate at the time of enrolment in the study. In addition, participants will have 4 telephone calls from an independent assessor to ask questions about their mental health (MADRS).

Participants will receive intranasal Esketamine 56mg or 84 mg once weekly for 4 weeks and 56 mg or 84 mg once every 2 weeks for 8 weeks as per Product Monograph

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have completed Study ZYL-730-01 through to Day 28
2. Adults aged 18-64
3. Participants must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign an informed consent.
4. Women must use a medically acceptable reliable means of contraception and must agree to use adequate birth control for the duration of the study and for 6 weeks after the last dose using methods from the permitted list for contraception.
5. If currently receiving medication for depression their antidepressant dose(s) must be stable for the previous 4 weeks prior to baseline.
6. Must be on a stable dose of all other medication(s) for at least 1-month prior to baseline visit., unless medication is to treat other short term conditions (i.e. influenza, upper respiratory track infections, pain, etc.)
7. Controlled hypertension and must be on a stable dose of antihypertensive medications for at least 3 months prior to the baseline visit.

Exclusion Criteria:

1. Women who plan to become pregnant, are pregnant or are breastfeeding.
2. Serious unstable medical illness, or any significant change in medical status at the baseline visit and during the study, as determined by the Investigator
3. Hormonal treatment (e.g., Estrogen) started within the 3 months prior to first dose of study treatment.
4. Participants who report treatment with a benzodiazepine, an opioid medication, or a mood stabilizer (such as valproic acid or lithium) at the baseline visit and within 2 weeks prior to the first dose of Esketamine .
5. Participants with confirmed psychotic disorder or symptoms, bipolar disorder and or clinically significant alcohol or substance misuse confirmed by a psychiatrist at the baseline visit. Those participants who develop symptoms of these may be withdrawn from the study, as determined by the Investigator
6. Current diagnosis of bulimia nervosa, or development of significant eating disorder symptoms at the baseline visit or during the study as determined by the Investigator
7. Participants who have been diagnosed with ADD/ADHD and who are also currently taking stimulant medication such as methylphenidate or another amphetamine-type medication, or who are diagnosed with this disorder or who start medication for this during the study.
8. Participants currently taking St John's Wort, Ginseng or Turmeric who start any of these during the study
9. Participants judged clinically to be actively at serious risk of self-harm or suicidal behaviour by the study team or psychiatrist at baseline or at any time during the study, as determined by the Investigator.
10. Blood pressure >140/90 at baseline
11. Participants who are unable to easily travel to the clinic for all of the in-person visits.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery Asberg Depression Rating Scale (MADRS) | Baseline, Day 26, 54 and 89
  The MADRS is a clinician rated 10-item scale where individuals score from 0-6 based on the severity of their symptoms with higher scores indicative of greater severity

SECONDARY OUTCOMES:
Change in Post-Traumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders (PCL-5 | Baseline, Day 26, 54 and 82
  A 20-item self-administered measure that assesses the presence and severity of PTSD symptoms derived from the symptoms of PTSD in DSM-5. Participants will be asked to rate how bothered they have been by each item in the 4 weeks on a 5-point Likert scale ranging from (0=Not at all to 4=Extremely). The PCL-5 is easily scored by summing all of the items for a total symptom severity score ranging between 0-80. Clinically meaningful PTSD symptoms are present if items are rated as a minimum of 2 = "Moderate" or higher.
Change in Patient Health Questionnaire (PHQ-9) | Baseline, Day 12, 26, 40, 54, 68 and 82
  A 9-item self-administered questionnaire to determine the presence and severity of depression which scores each of the 9 DSM-IV criteria as "0"(not at all), to "3" (nearly everyday
Change in Generalized Anxiety Disorder Questionnaire (GAD-7) | Baseline, Day 12, 26, 40, 54, 68 and 82
  A 7-item self-administered questionnaire to measure the severity of the levels of anxiety. Each item can be scored 0-3, giving a total score of 0-21.
Change in Rosenberg Self-Esteem Questionnaire (RSES) | Baseline, Day 26, 54 and 82
  A 10-item self administered questionnaire to measure change in self esteem following psychological intervention. Each item scoring from 1-4, and higher scores indication greater self-esteem
Change in Quality of Life 8 Dimensional Questionnaire (AQoL-8D) | Baseline, Day 26, 54 and 82
  Self administered questionnaire measuring quality of life across 8 domains: independent living, happiness, mental health, coping, relationships, self-worth, pain and senses

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Chue, MBBCh, Principal Investigator — Amygdala Associates Inc.

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available to other members of the study team including Dr. Craig Buchholz
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Throughout the study
Access Criteria: Involved in data collection